CLINICAL TRIAL: NCT07211100
Title: Evaluation of the Impact of a Mobile Application Developed for Hemodialysis Patients on Treatment Adherence, Symptom Management and Clinical Parameters.
Brief Title: Evaluation of the Effectiveness of a Mobile Application Developed for Hemodialysis Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, İlknur Palaz, Doctoral Student and lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBU-GHEM-IP-01
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: End-Stage Renal Disease Requiring Haemodialysis; Mobile Application
Keywords: hemodialiysis; mobile application; mobil health; pain; fatigue; itching; nursingcare; adaptation; esrd
MeSH Terms: conditions — Pain; Fatigue; Pruritus; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups: an intervention group and a control group. The intervention group will use the mobile health application developed by the research team, while the control group will receive standard care without the application. Both groups will be followed simultaneously, and outcomes will be measured at baseline (T0), 1 month (T1), and 2 months (T2). Block randomization will be used to ensure balanced group allocation.
Who Masked: Outcomes Assessor
Masking Description: No additional parties are masked other than the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Intervention Arm (Experimental): Participants assigned to this arm will receive the mobile health application developed by the research team. The application includes modules on treatment adherence (medication, diet, fluid restriction, dialysis attendance), symptom management (fatigue, pain, itching), nutrition guidance, exercise recommendations, reminder notifications, expert Q&A, and personal tracking.
  Interventions: Behavioral: Mobile Health Application
- Arm 2 - Control Arm (No Intervention): Participants in this group will receive standard hemodialysis care without the mobile application. Standard care includes routine clinical follow-up, medical treatment, and nursing care provided at the dialysis center.

INTERVENTIONS:
Behavioral: Mobile Health Application — A mobile health application developed by the research team to support hemodialysis patients. The application includes modules on treatment adherence (medication, diet, fluid restriction, dialysis attendance), symptom management (fatigue, pain, itching), nutrition guidance, exercise recommendations, reminder notifications, expert Q&A, and personal tracking. The aim is to improve adherence to treatment, reduce symptom burden, and support patient self-care.
  Arms: Arm 1 - Intervention Arm

SUMMARY:
This study aims to evaluate the effectiveness of a mobile health application developed for adult patients undergoing hemodialysis treatment. The mobile application includes modules on adherence to medication, diet, and fluid restrictions, symptom management (fatigue, pain, itching), nutrition guidance, exercise recommendations, and motivational content. It also features reminder notifications, an "Ask the Expert" module, and personal symptom tracking.

The research will be conducted as a single-center, single-blind, randomized controlled experimental study. Participants will be assigned to intervention and control groups using block randomization. The intervention group will receive the mobile application, while the control group will receive standard care. Assessments will be carried out at baseline (T0), 1st month (T1), and 2nd month (T2).

The measurement tools to be used include the End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ), Post-Dialysis Fatigue Scale, 5-D Itch Scale, Visual Analog Scale (VAS) for pain, and the Mobile Application Usability Scale. In addition, clinical parameters such as serum potassium, phosphorus, and albumin will be evaluated.

A total of 72 patients (36 intervention, 36 control) will be included in the study. This study aims to assess the impact of a mobile health application on treatment adherence, symptom management, and clinical parameters among hemodialysis patients, and to develop a digital health model that can be integrated into nursing care.

DETAILED DESCRIPTION:
Chronic kidney disease is a major global public health problem, and most patients with end-stage renal disease (ESRD) depend on hemodialysis to survive. Patients undergoing hemodialysis often experience difficulties with treatment adherence, challenges related to dietary and fluid restrictions, as well as common symptoms such as fatigue, pain, and itching. These problems negatively affect their quality of life. Previous studies have reported that more than half of hemodialysis patients demonstrate poor treatment adherence, which is associated with increased mortality. Therefore, innovative and technology-based approaches are needed to improve adherence and reduce symptom burden.

In recent years, mobile health (mHealth) applications have been increasingly used in the management of chronic diseases. Such applications enable patients to monitor their health more closely, improve medication and dietary adherence, and receive support for symptom management. However, most existing studies in the literature have focused on only one dimension of adherence (such as medication or diet) and have not comprehensively evaluated symptom management together with biochemical parameters.

This study aims to investigate the effect of a newly developed mobile health application, created by the research team, on treatment adherence, symptom management (fatigue, pain, itching), and clinical parameters (serum potassium, phosphorus, albumin) among hemodialysis patients. The study will be conducted as a single-center, single-blind, randomized controlled trial including a total of 72 patients (36 intervention, 36 control). Participants will be assigned to groups using block randomization. The intervention group will receive the mobile application, while the control group will continue with standard care.

The mobile application has been specifically designed and developed by the research team to meet the needs of hemodialysis patients. It consists of modules on treatment adherence (medication, diet, fluid restriction, dialysis attendance), symptom management (fatigue, itching, pain), nutrition guidance, exercise recommendations, reminder notifications, a question-answer section with experts, and personal monitoring. The aim is to improve patients' self-care abilities and reduce their symptom burden.

Data will be collected at baseline (T0), 1st month (T1), and 2nd month (T2). Measurement tools include the End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ), Post-Dialysis Fatigue Scale, 5-D Itch Scale, Visual Analog Scale (VAS) for pain, and the Mobile Application Usability Scale. In addition, laboratory parameters such as serum potassium, phosphorus, and albumin will be evaluated.

At the end of the study, scientific evidence will be obtained regarding whether the mobile health application developed by the research team is effective in improving treatment adherence, alleviating symptoms, and enhancing clinical outcomes in hemodialysis patients. The findings are expected to provide a model for integrating digital health applications into nursing care and to contribute to the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosed with end-stage renal disease (ESRD).
* Receiving maintenance hemodialysis treatment for at least 3 months.
* Able to use a smartphone and willing to install the mobile health application.
* Voluntarily agreeing to participate in the study and providing written informed consent.

Exclusion Criteria:

* Patients with cognitive impairment, severe psychiatric disorders, or communication barriers that may interfere with participation.
* Patients with visual or hearing impairments that prevent the use of the mobile application.
* Patients who have undergone kidney transplantation or are scheduled for transplantation within the study period.
* Patients with serious comorbid conditions requiring hospitalization (e.g., advanced cancer, severe heart failure).
* Participation in another interventional clinical trial within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Treatment Adherence Score | Baseline (T0), 1 month (T1), and 2 months (T2).
  Treatment adherence will be assessed using the End-Stage Renal Disease Adherence Questionnaire (ESRD-AQ). Higher scores indicate better adherence. The intervention group will use the mobile health application, while the control group will receive standard care.
Change in Symptom Burden | Baseline (T0), 1st month (T1), and 2nd month (T2).
  ymptom burden will be evaluated using the Edmonton Symptom Assessment Scale (ESAS), which covers multiple symptoms such as fatigue, itching, pain, sleep disturbance, and other common hemodialysis-related complaints. Higher scores reflect higher symptom severity.

SECONDARY OUTCOMES:
Mobile Application Usability | At the 2nd month and after.
  Measured by the Mobile Application Usability Scale among intervention group participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane State Hospital, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is a doctoral thesis project, and data use is restricted to the research team in accordance with ethics committee approval.